CLINICAL TRIAL: NCT02199080
Title: Etude du Dosage Des d-dimères sériques Pour le Diagnostic d'Exclusion Des Thrombi Intra-atriaux Avant Ablation Endocavitaire de Fibrillation Atriale
Brief Title: D-dimer Assay for the Exclusion of Intra-atrial Thrombus Risk Before Ablation of Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe Hospitalier de la Rochelle Ré Aunis (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014/P02/001; 2013-A01700-45 (Other: French National Agency for Medicines/Health Products Safety)
Record Dates: First submitted 2014-07-22; First posted 2014-07-24 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Atrial fibrillation (Other): D-dimer assay before ablation of atrial fibrillation
  Interventions: Other: D-dimer assay before ablation of atrial fibrillation

INTERVENTIONS:
Other: D-dimer assay before ablation of atrial fibrillation — Blood sample collection for D-dimers measurement

SUMMARY:
The purpose of this study is to determine whether D-dimer dosage allow to exclude risk of intraatrial thrombus before performing an ablation of atrial fibrillation

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years.
* Patients hospitalized for ablation of atrial fibrillation or symptomatic left flutter
* Patient informed of the study

Exclusion Criteria:

* Age <18 years.
* Patients under guardianship
* Pregnant woman
* Contraindication to transesophageal echocardiography
* transesophageal echocardiography made in another center as the center of ablation
* Refusal of the patient to participate in the study
* Patient participating in another interventional study in which an intervention related to biomedical research is performed before the transesophageal echocardiography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2506 (Actual)
Dates: Start 2014-07-28; Primary Completion 2016-01 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antoine MILHEM, MD, Principal Investigator — Groupe Hospitalier de la Rochelle Ré Aunis
Locations (37):
- France (37):
  - Service de cardiologie, CH de la Région d'Annecy, Annecy
  - Centre Hospitalier d' Auxerre, Auxerre
  - Service de cardiologie, CH Avignon, Avignon
  - Clinique La Fourcade, Bayonne
  - Service de cardiologie, CHU Bordeaux, Bordeaux
  - Service de cardiologie, CHU Brest, Brest
  - Service de cardiologie, CHU Caen, Caen
  - Service de cardiologie, CHU Clermont Ferrand, Clermont-Ferrand
  - Service de cardiologie, AP Hôpital Henri Mondor, Créteil
  - Service de cardiologie, CHU Dijon, Dijon
  - Groupe Hospitalier de la Rochelle Ré Aunis, La Rochelle
  - Service de cardiologie, CH Le Mans, Le Mans
  - Service de cardiologie, CHU Limoges, Limoges
  - Service de cardiologie, HCL Groupement Est, Lyon
  - Service de cardiologie, APM Hôpital de La Timone, Marseille
  - Service de cardiologie, CHI Aix Pertuis CHPA-CHIAP, Marseille
  - Service de cardiologie, Hôpital Saint Joseph, Marseille
  - Service de cardiologie, Institut Jacques Cartier, Massy
  - Service de cardiologie, CHR Metz Thionville, Metz
  - Service de cardiologie, CHI Le Raincy Montfermeil, Montfermeil
  - Service de cardiologie, CHU Nancy, Nancy
  - Service de cardiologie, Nouvelles Cliniques Nantaises, Nantes
  - Service de cardiologie, CHU Nîmes, Nîmes
  - Service de cardiologie, HP Les Franciscaines, Nîmes
  - Service de cardiologie, AP Hôpital la Pitié Salpêtrière, Paris
  - Service de cardiologie, Groupe Hospitalier Bichat Claude Bernard, Paris
  - Service de cardiologie, Institut Mutualiste Montsouris, Paris
  - Service de cardiologie, CH Pau, Pau
  - Service de cardiologie, CHU Poitiers, Poitiers
  - Service de cardiologie, CHU Rennes, Rennes
  - Service de cardiologie, CHU Rouen, Rouen
  - Service de cardiologie, Centre Cardiologique du Nord, Saint-Denis
  - Service de cardiologie, CHU Saint Etienne, Saint-Etienne
  - Service de cardiologie, CHU Toulouse Hôtel Dieu St Jacques, Toulouse
  - Service de cardiologie, Clinique Saint Gatien, Tours
  - Service de cardiologie, Clinique Saint Joseph, Trélaze
  - Service de cardiologie, Polyclinique Vauban, Valenciennes

REFERENCES:
- [Result] Milhem A, Ingrand P, Treguer F, Cesari O, Da Costa A, Pavin D, Rivat P, Badenco N, Abbey S, Zannad N, Winum PF, Mansourati J, Maury P, Bader H, Savoure A, Sacher F, Andronache M, Allix-Beguec C, De Chillou C, Anselme F; ATE Study Group. Exclusion of Intra-Atrial Thrombus Diagnosis Using D-Dimer Assay Before Catheter Ablation of Atrial Fibrillation. JACC Clin Electrophysiol. 2019 Feb;5(2):223-230. doi: 10.1016/j.jacep.2018.09.009. Epub 2018 Nov 1. PMID 30784695

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Atrial Fibrillation
Started | 2506
Completed | 2494
Not Completed | 12
Not completed — Protocol Violation | 12

BASELINE CHARACTERISTICS:
Arm/Group | Atrial Fibrillation
Number analyzed (Participants) | 2494
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 676
  Male | 1818
Region of Enrollment [Number; unit: participants]
  France | 2494
Paroxysmal fibrillation [Count of Participants; unit: Participants] | 1335
Persistent fibrillation [Count of Participants; unit: Participants] | 996
Left atrial tachycardia [Count of Participants; unit: Participants] | 163
left ventricular ejection fraction [Mean (Standard Deviation); unit: percentage of ejection fraction] | 57.4 (10.0)
Medical history [Count of Participants; unit: Participants]
  Previous left atrial ablation | 593
  Hypertension | 916
  Diabetes mellitus | 227
  Heart failure | 304
  Stroke | 115
  Venous thromboembolism | 45
  Inflammatory disease | 34
  Neoplasia | 25
  Infectious disease | 6
  Recent surgery | 4
Anticoagulation [Count of Participants; unit: Participants]
  No anticoagulant therapy | 235
  DABIGATRAN | 269
  RIVAROXABAN | 596
  APIXABAN | 321
  Effective Vitamin K antagonists | 814
  Non effective Vitamin K antagonists | 245
  Other | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Atrial Thrombus Diagnosed by Transoesophageal Ultrasound
Time Frame: up to 48 hours before ablation
Measure: Count of Participants; unit: Participants
Arm/Group | Atrial Fibrillation
Number analyzed (Participants) | 2494
Participants | 48

2. Secondary Outcome: CHADS2 Score
Description: CHADS2 score (congestive heart failure=1, hypertension=1, diabetes mellitus=1, history of stroke or transient ischemic attack=1, and age under 75=1)
Time Frame: 48 hours before ablation
Measure: Count of Participants; unit: Participants
Groups:
- Atrial Thrombus: Patients with atrial thrombus diagnosed by pre-procedural transoesophageal echocardiography
- No Atrial Thrombus: Patients with no atrial thrombus diagnosed by pre-procedural transoesophageal echocardiography
Arm/Group | Atrial Thrombus | No Atrial Thrombus
Number analyzed (Participants) | 48 | 2446
Participants
  CHADS2 score = 0 | 5 | 1277
  CHADS2 score = 1 | 20 | 744
  CHADS2 score = 2 | 13 | 299
  CHADS2 score ≥ 3 | 10 | 126

3. Secondary Outcome: Risk Factors
Description: variables related to the presence of atrial thrombus
Time Frame: 48 hours before ablation
Measure: Count of Participants; unit: Participants
Arm/Group | Atrial Thrombus | No Atrial Thrombus
Number analyzed (Participants) | 48 | 2446
Participants
  Age (≥ 75yrs) | 8 | 148
  Female gender | 15 | 661
  Persistent fibrillation | 28 | 968
  Hypertension | 30 | 886
  Diabetes mellitus | 9 | 218
  Heart failure | 19 | 285
  History of stroke | 6 | 109
  Previous left atrial ablation | 9 | 584
  Anticoagulation prior to ablation | 47 | 2212

4. Secondary Outcome: Atrial Thrombus Exclusion (ATE) Score
Description: The following thromboembolic risk factors mark 1 point if present in patient:
  * hypertension = 1 point
  * cardiac insufficiency = 1 point
  * history of stoke = 1 point
  * d-dimer level >270ng/mL = 1 point The sum corresponds to the ATE score
Time Frame: 48 hours before ablation
Measure: Count of Participants; unit: Participants
Arm/Group | Atrial Thrombus | No Atrial Thrombus
Number analyzed (Participants) | 48 | 2446
Participants
  ATE score = 0 | 0 | 911
  ATE score = 1 | 23 | 965
  ATE score = 2 | 14 | 467
  ATE score = 3 | 10 | 101
  ATE score = 4 | 1 | 2

ADVERSE EVENTS:
Time Frame: Serious and non-serious adverse events (biological and clinical) that occured between the signature of the consent and the end of patient participation were reported. The duration of patient participation was 48 hours.
Arm/Group | Atrial Fibrillation
All-Cause Mortality (participants affected / at risk) | 0/2506
Serious Adverse Events (participants affected / at risk) | 0/2506
Other Adverse Events (participants affected / at risk) | 0/2506

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No